CLINICAL TRIAL: NCT06644651
Title: Prospective Associations of Pericoronary Adipose Tissue Computed Tomography Attenuation With Coronary Plaque Features and Major Adverse Cardiovascular Events in a Population With Diabetes Mellitus
Brief Title: Fat Around Heart Arteries as a Measure of Inflammation in Patients With Diabetes
Acronym: PCAT-DM
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PCAT-DM
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Atherosclerosis, Coronary; Diabetes Mellitus; Diabetes Mellitus Type 2; Inflammation; Inflammation Plaque, Atherosclerotic; Perivascular Disease
Keywords: Atherosclerotic Plaque; Coronary artery disease; Atherosclerosis, coronary; Inflammation; Pericoronary adipose tissue; Coronary inflammation; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Diabetes Mellitus, Type 2; Inflammation; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting blood samples at baseline and at 12 months follow-up within one week from the day of the CCTA.
  Biochemistry included; HbA1c, low-density lipoprotein (LDL), high-density lipoprotein HDL, triglycerides (TG), creatinine, high-sensitivity C-reactive peptide (hs-CRP), high-sensitivity Troponine T (hs-TNT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes mellitus: The study population consists of participants with type 2 diabetes mellitus who are cardiac asymptomatic and have no known coronary heart disease. Participants underwent a baseline examination and CCTA scan, followed by a 12-month visit with repeated examinations and a second CCTA scan. A journal audit will be conducted for all participants approximately 7 years after the baseline CCTA scan.

SUMMARY:
In this prospective study, the objective is to investigate inflammation in the arteries of the heart. A heart CT scan (CCTA) will be used to measure inflammation by assessing the fat tissue surrounding the arteries of the heart. Participants with type 2 diabetes who have no heart symptoms have been examined, using a CCTA at the start of the study and again after 12 months.

This study aims to answer the following questions:

* Can inflammation in the surrounding fat tissue at the baseline CCTA predict the amount and type of plaque, and the presence of harmful plaque characteristics present after 12 months? (paper 1)
* Do changes in inflammation in the surrounding fat tissue from baseline to the 12 months CCTA correlate with the amount and type of plaque and the presence of harmful plaque characteristics at the 12 months CCTA? (paper 1)
* Is inflammation in the surrounding fat tissue a predictor for the development of cardiovascular events after a follow-up period of 7 years? (paper 2)
* Do changes in inflammation in the surrounding fat tissue after 12 months predict the later development of cardiovascular events after a follow-up period of 7 years? (paper 2)

DETAILED DESCRIPTION:
Background and significance:

Inflammation in the coronary arteries plays a significant role in the development of heart disease, particularly in individuals with type 2 diabetes (T2D), who are at an increased risk. However, this inflammation has been difficult to detect because the currently used biomarkers have limited accuracy in identifying inflammation in the coronary arteries.

Exiting advancements have been made in the field of coronary CT angiography (CCTA). CCTA enables the measurement of the pericoronary adipose tissue (PCAT) attenuation, which refers to the fat tissue surrounding the coronary arteries. PCAT and the coronary arteries have a bidirectional communication, and when PCAT is exposed to high inflammation it causes the fat-structure to change. These structural changes in PCAT can be detected with a CCTA scan. Additionally, a CCTA scan can assess plaque characteristics, such as the amount of plaque (burden), the type of plaque (composition), and the presence of high-risk plaque features, all of which, are linked to major adverse cardiovascular events (MACE). Furthermore, recent studies have shown that PCAT attenuation can predict cardiac events and mortality.

The PCAT-DM study is a post-hoc analysis from the CARPE-DM study (NCT03016910). The goal of this prospective study is to investigate whether PCAT attenuation and/or PCAT changes are associated with high-risk plaque features, plaque composition and burden. Additionally, the study aims to investigate whether PCAT attenuation and/or PCAT changes can predict development of MACE over a follow-up period of 7 years.

Setting and study population:

A single-center prospective observational study at Odense University Hospital, Svendborg, Denmark. The study enrollment began in March 2016 and ended in September 2017. The study population consists of cardiovascularly asymptomatic participants with type 2 diabetes mellitus.

Examinations:

A total of 314 patients were examined with a CCTA scan at baseline and again after 12 months. The following examinations were conducted at baseline:

* CCTA scan
* CAC-score
* Blood pressure and pulse frequency
* Height, weight, waist to hip-ratio
* Blood samples and urin samples
* Medical history After 12 months, all of the above examinations were repeated.

Journal audits will be performed in the period from September 2024 to January 2025 to examine the number of clinical events according to the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Capable of giving written informed consent
* Type 2 diabetes mellitus

Exclusion Criteria:

* History of CAD
* Symtoms of CAD (angina)
* Any tachyarrhythmias making CCTA impossible
* Estimated glomerular filtration rate (eGFR) under 45 ml/min
* Allergy to iodine contrast
* Critical illness with life expectancy less than 1 year
* Documented heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes who were cardiac asymptomatic and had no history of CAD. Participants were recruited from the Endocrinology Outpatient Clinic and the Retina Photographhy Clinic at Odense University Hospital, Svendborg, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2025-02 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Baseline PCAT attenuation and plaque features at the 12-month CCTA | 12 months
  Cardiac assessments at the 12-month CCTA scan include:
  Plaque composition, measured by the volume of different plaque types. Plaque burden is measured as compositional plaque volume adjusted by vessel length (normalized atheroma volume).
  High-risk plaque features assessed include positive remodeling (PR), low-attenuated plaque (LAP), napkin-ring sign (NRS), and spotty calcifications (SC).
Changes in PCAT attenuation and plaque features at the 12-month CCTA | 12 months
  Changes in PCAT attenuation from baseline to the 12-month CCTA will be measured.
  Cardiac assessments at the 12-month CCTA scan include:
  Plaque composition, measured by the volume of different plaque types. Plaque burden is measured as compositional plaque volume adjusted by vessel length (normalized atheroma volume). High-risk plaque features assessed include positive remodeling (PR), low-attenuated plaque (LAP), napkin-ring sign (NRS), and spotty calcifications (SC).
Baseline PCAT attenuation and MACE | 7 years
  Baseline PCAT attenuation will be used to predict major adverse cardiovascular (CV) events (MACE), including CV death, non-fatal acute myocardial infarction (AMI), non-fatal stroke, heart failure (HF) de novo, and hospitalization for HF, over a 7-year period following the CCTA scan.
Changes in PCAT attenuation after 12-month and MACE | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict major adverse cardiovascular (CV) events (MACE), including CV death, non-fatal acute myocardial infarction (AMI), non-fatal stroke, heart failure (HF) de novo, and hospitalization for HF, over a 7-year period following the CCTA scan.

SECONDARY OUTCOMES:
PCAT attenuation and de novo heart failure | 7 years
  Baseline PCAT attenuation will be used to predict de novo heart failure over a 7-year period following the CCTA scan.
PCAT attenuation and non-fatal acute myocardial infarction | 7 years
  Baseline PCAT attenuation will be used to predict non-fatal acute myocardial infarction (AMI) over a 7-year period following the CCTA scan.
PCAT attenuation and non-fatal stroke | 7 years
  Baseline PCAT attenuation will be used to predict non-fatal stroke over a 7-year period following the CCTA scan.
PCAT attenuation and hospitalization for HF | 7 years
  Baseline PCAT attenuation will be used to predict hospitalization for heart failure (HF) over a 7-year period following the CCTA scan.
PCAT attenuation and CV death | 7 years
  Baseline PCAT attenuation will be used to predict cardiovascular (CV) death over a 7-year period following the CCTA scan.
PCAT attenuation and PAD | 7 years
  Baseline PCAT attenuation will be used to predict peripheral artery disease (PAD) over a 7-year period following the CCTA scan.
PCAT attenuation and CV revascularization | 7 years
  Baseline PCAT attenuation will be used to predict CV (cardiovascular) revascularization over a 7-year period following the CCTA scan.
PCAT attenuation and all-cause mortality | 7 years
  Baseline PCAT attenuation will be used to predict all-cause mortality over a 7-year period following the CCTA scan.
Changes in PCAT attenuation and non-fatal acute myocardial infarction | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict non-fatal acute myocardial infarction (AMI) over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and hospitalization for HF | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict hospitalization for heart failure (HF) over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and non-fatal stroke | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict non-fatal stroke over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and PAD | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict peripheral artery diasease (PAD) over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and CV death | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict cardiovascular (CV) death over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and CV revascularization | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict cardiovascular (CV) revascularization over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and all-cause mortality | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict all-cause mortality, over a 7-year period following the baseline CCTA scan.
Changes in PCAT attenuation and de novo heart failure | 7 years
  Changes in PCAT attenuation from baseline to the 12-month CCTA scan will be used to predict de novo heart failure (HF) over a 7-year period following the baseline CCTA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Professor, Principal Investigator — Odense University Hospital - Svendborg
Locations (1):
- Cardiovascular Research Unit, Svendborg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Overgaard KS, Andersen TR, Heinsen LJ, Pararajasingam G, Mohamed RA, Madsen FS, Biesenbach IIA, Hojlund K, Lambrechtsen J, Auscher S, Egstrup K. Pericoronary adipose tissue attenuation predicts compositional plaque changes: a 12-month longitudinal study in individuals with type 2 diabetes without symptoms or known coronary artery disease. Cardiovasc Diabetol. 2025 Mar 28;24(1):143. doi: 10.1186/s12933-025-02694-9. PMID 40155929